CLINICAL TRIAL: NCT04959435
Title: Understanding the Role of the Salivary Microbiota and Microbiota Associated to Mucosa in Behçet's Disease
Brief Title: Understanding the Role of Oral Microbiota in Behçet's Disease (BEHCETBIOT)
Acronym: BEHCETBIOT
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RBHP 2021 ANDRE; 2021-A01648-33 (Other: ANSM)
Record Dates: First submitted 2021-07-02; First posted 2021-07-13 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Behçet Disease; Physiopathology; Microbiota; Oral Microbiota
MeSH Terms: conditions — Behcet Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Behcet's disease patients
  Interventions: Other: biological samples collection
- Controls: Controls that matched two to two at case according to sex,social status and diet.
  Interventions: Other: biological samples collection

INTERVENTIONS:
Other: biological samples collection — samples of blood, faeces, saliva, dental plaque, oral mucosa, genital mucosa

SUMMARY:
Behçet's disease (BD) is a systemic vasculitis that affects, especially, young people.

Although its etiology remains unexplained, data suggest that the inflammatory response during BD results from a disruption of the homeostasis of innate and adaptive immune responses in genetically predisposed people. The microbiota could play a triggering role in BD, in particular the salivary and dental plaque microbiota. The aim of the Behçetbiot study is therefore to establish microbial profiles of dental plaque, pathological (on the mouth ulcer) and non-pathological mucous membrane, salivary and digestive and to compare them with control subjects not suffering from BD, related to the first degree, of the same socio-cultural level and to determine whether dysbiosis is correlated with a local and systemic pro-inflammatory response, by measuring salivary level of pro-inflammatory cytokines and blood level of CRP, fibrinogen, orosomucoïd and haptoglobin, and to compare them with controls.

DETAILED DESCRIPTION:
All patients and their controls are sampled for stool, saliva, dantal plaque, oral mucosa, genital mucosa and blood during an annual follow-up visit or if they are hospitalised.

Plaque, oral mucosa, genital mucosa salivary and blood will be collected during an annual follow-up visit.

For stool samples, the collection material will be provided to the patient and they will be able to take the sample at home and bring it to the clinic, or send them via a carrier within 3 days.

All the samples related to the study will be taken in the internal medicine in Clermont-Ferrand (France) or Pitie Salpêtrière, department of internal medecine, Paris,France or ophthalmology departments in Clermont-Ferrand.

All sample will be stocked in biological center in Clermont-Ferrand before analyze.

Microbiota analyzes will be realise at M2iSH laboratoty, inflammatory cytokines will be analyze in Clermont-Ferrand immunology laboratory, and pro-inflammatory parameters will be analyse in biochimy laboratory in Clermont-Ferrand.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet the International criteria for the classification of Behçet's disease, revised in 2013)
* Patient who had developed the disease in the 5 years preceding the study.

Exclusion Criteria:

* Pregnant or breastfeeding women, or women who may be pregnant or breastfeeding.
* Subject placed under judicial protection.
* Patient had received antibiotic or probiotic or symbiotic therapy in the 6 weeks preceding inclusion

Ages: 18 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: Patient who have behçet's disease.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
Oral microbiota | Day 0
  Establish microbial profiles (quantitative and qualitative via analysis of bacterial DNA sequences encoding 16S rRNA) of dental plaque, pathological (on the aphta) and non-pathological oral mucosa and and salivary and compared them to control without Behçet's disease matched for sex, diet and socio-cultural level.

SECONDARY OUTCOMES:
Intestinal microbiota | Day 0
  Establish microbial profiles (quantitative and qualitative via analysis of DNA sequences encoding 16S rRNA) of the intestinal microbiota by studying feces and comparing them to controls without Behçet's disease, of the same sex, diet and socio-cultural level
Short fatty acid | Day 0
  Determination of short-chain fatty acids (HPLC technique) in the stools of Behçet patients and compare them to control patients without Behçet's disease, of the same sex, diet and socio-cultural level
Pro-inflammatory cytokines | Day 0
  Determination of blood and saliva levels of IL-1beta, IL-6, IL-17, IL21, IL-23, Il-10, IFN gamma and TNF alpha (ELISA technique or multiplexed assay) and compare them to patients without Behçet disease, of the same sex, diet and socio-cultural level.
  socio-cultural level
genital microbiota | Day 0
  Establish microbial profiles (quantitative and qualitative via analysis of DNA sequences encoding 16S rRNA) of the intestinal microbiota by studying feces and comparing them to controls without Behçet's disease, of the same sex, diet and socio-cultural level

CONTACTS AND LOCATIONS:
Overall Officials: Marc André, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (2):
- France (2):
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - Hopital La Pitié Salpetriere, Paris

IPD SHARING:
Plan to Share IPD: No
Data are reserved for M2ISH laboratory team .